CLINICAL TRIAL: NCT01812304
Title: Objective Structured Assessment of Technical Skills Evaluation of Theoretical Compared With hands-on Training of Shoulder Dystocia Management: a Randomized Controlled Trial.
Brief Title: Theoretical Compared With hands-on Training of Vaginal Breech Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Dr. med. Clemens Tempfer, MBA, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VB-01
Record Dates: First submitted 2013-03-08; First posted 2013-03-18 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Vaginal Abnormality - Baby Delivered

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hands-on training (Experimental): probands perform predefined maneuvers to manage a vaginal breech hands-on after one instruction
  Interventions: Other: hands-on training
- frontal teaching (Active Comparator): Probands perform predefined maneuvers to resolve a vaginal breech after forntal teaching
  Interventions: Other: frontal teaching

INTERVENTIONS:
Other: hands-on training — the intervention consists of a predefined hands-on training program including 25 technical steps to manage a vaginal breech
  Arms: hands-on training
Other: frontal teaching — one teacher demonstrates all 25 items listed in the OSATS checklist. Probands listen and watch.
  Arms: frontal teaching

SUMMARY:
This trial aims to assess the hypothesis that hands-on training of vaginal breech delivery on a pelvic model is significantly better in terms of a technical skills scoring system compared to frontal teaching.

DETAILED DESCRIPTION:
Primary endpoint is a score describing technical proficiency, ie the OSATS score, consisting of 25 items. Each item, if done correctly, is awarded one point. The maximum OSATS score is 25.

Secondary endpoints are performance time in seconds, cinfidence using a scale from 1-5 with one being very confident and 5 having no confidence when performing the procedures, and self-assessment using a scale of 1-5 with 1 being the optimal grade.

This is a two-arm study. The experimental arm uses a hands-on training and the control arm a frontal teaching approach. The allocation is randomized and single-blinded.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* able to understand German
* Medical student

Exclusion criteria:

* significant language barrier
* previous experience with vaginal breech training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
OSATS Score | probands are tested after training within an hour
  OSATS Scores are assessed on a pelvic model by a blinded assessor immediately after training (1 arm hands-on, 1 arm forntal teaching)

SECONDARY OUTCOMES:
OSATS Scores | 72 Hours after training
  identical to primary outcome, but 72 hours later

OTHER OUTCOMES:
confidence, speed, self assessment | immediately after training and 72 hours later

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Tempfer, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Buerkle B, Rueter K, Hefler LA, Tempfer-Bentz EK, Tempfer CB. Objective Structured Assessment of Technical Skills (OSATS) evaluation of theoretical versus hands-on training of vaginal breech delivery management: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):252-6. doi: 10.1016/j.ejogrb.2013.09.015. Epub 2013 Sep 25. PMID 24103530